CLINICAL TRIAL: NCT03382379
Title: Transcranial Direct Current Stimulation to Modulate Top-Down Regulation for Drug Craving in Methamphetamine Use Disorder (MUD)
Brief Title: Transcranial Direct Current Stimulation to Modulate Top-Down Regulation for Drug Craving in Methamphetamine Use Disorder
Acronym: NeuroMethDC
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Laureate Institute for Brain Research, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 2017-005-00
Record Dates: First submitted 2017-12-01; First posted 2017-12-22 (Actual); Last update posted 2019-06-07 (Actual); Status verified 2019-03

CONDITIONS: Amphetamine Use Disorders
Keywords: methamphetamine; transcranial Direct Current Stimulation; functional Magnetic Resonance Imaging; amphetamine; drug craving

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active (Experimental): Participants in the active arm will receive 2 milliamp anodal transcranial Direct Current Stimulation (tDCS) over the Dorso-Lateral Pre-Frontal Cortex (DLPFC).
  Interventions: Device: Active transcranial Direct Current Stimulation (tDCS)
- Sham (Placebo Comparator): Participants in the Sham arm will receive sham transcranial Direct Current Stimulation (tDCS) over the Dorso-Lateral Pre-Frontal Cortex (DLPFC).
  Interventions: Device: Sham transcranial Direct Current Stimulation (tDCS)

INTERVENTIONS:
Device: Active transcranial Direct Current Stimulation (tDCS) — Transcranial Direct Current Stimulation (tDCS) as a device-based technology is employed by applying a very weak (2 mAmp) direct current over the skull for 1200 seconds with 30 seconds ramp up to 2 mAmp, and 30 seconds ramp down at the end.
  Arms: Active
Device: Sham transcranial Direct Current Stimulation (tDCS) — Sham Transcranial Direct Current Stimulation (tDCS) as a device-based technology is employed by applying a very weak direct current over the skull. Sham mode will have just 30 seconds ramp up to 2 mAmp, 40 seconds on 2 mAmp stimulation and, 30 seconds ramp down with 1160 seconds no stimulation (just impedance control).
  Arms: Sham

SUMMARY:
Methamphetamine use disorder (MUD) is among the costliest and deadliest substance use disorders (SUDs) world-wide and is frequently comorbid with other mental health conditions. There is no empirically validated medical treatment for MUD. Drug craving is the signature aspect of MUD and other substance use disorders and has been associated with continued drug use and relapse. The investigators and others have shown that transcranial direct current stimulation (tDCS) over dorsolateral prefrontal cortex (DLPFC) can modulate drug craving in different SUDs. tDCS is a method of non-invasive brain stimulation and is a low-cost scalable technology without any serious side effects that delivers low levels of direct current (0.1-2 mAmp) transcranially. However, there are significant inter-individual differences in response to tDCS, which is not well understood but can have profound impact on efficacy. Meanwhile, there are no studies with neuroimaging to show how tDCS affects drug craving. Investigators propose the first combined tDCS/functional Magnetic Resonance Imaging (fMRI) study to examine the acute effects of tDCS on neural substrates underlying drug induced craving.

DETAILED DESCRIPTION:
Methamphetamine use disorder (MUD) is among the costliest and deadliest substance use disorders (SUDs) world-wide and is frequently comorbid with other mental health conditions. There is no empirically validated medical treatment for MUD. Drug craving is the signature aspect of MUD and other substance use disorders and has been associated with continued drug use and relapse. The investigators and others have shown that transcranial direct current stimulation (tDCS) over dorsolateral prefrontal cortex (DLPFC) can modulate drug craving in different SUDs. tDCS is a method of non-invasive brain stimulation and is a low-cost scalable technology without any serious side effects that delivers low levels of direct current (0.1-2 mAmp) transcranially. However, there are significant inter-individual differences in response to tDCS, which is not well understood but can have profound impact on efficacy. Meanwhile, there are no studies with neuroimaging to show how tDCS affects drug craving. The investigators propose the first combined tDCS/functional Magnetic Resonance Imaging (fMRI) study to examine the acute effects of tDCS on neural substrates underlying drug induced craving. The investigators hypothesize that tDCS amplifies DLPFC's top-down modulatory role via its connectivity to other cortical-subcortical areas. In this double blind randomized experimental design, the investigators will recruit 60 people with MUD during their early abstinence phases into parallel arms with active and sham DLPFC tDCS. Each subject will undergo resting state and task based (drug cue exposure paradigm) functional MRI pre and post tDCS. The investigators will conduct individual difference analyses to explore the potential predictors for tDCS response, including pre-tDCS top-down connectivity measures of DLPFC and other subjective, clinical, behavioral, structural, and functional variables. The results of this study will provide neuroscience-based evidence for the efficacy of tDCS and will advance the field towards precision addiction medicine.

ELIGIBILITY:
Inclusion Criteria:

1. English speaking.
2. Diagnosed with Methamphetamine Use Disorder (last 12 months) based on the Mini International Neuropsychiatric Interview (MINI) interview (Diagnostic and Statistical Manual of Mental Disorders-DSM-5)
3. Being abstinent from methamphetamine in an addiction treatment program for at least one week based on medical records or self-report
4. Positive response to Methamphetamine cue-reactivity screening (MCS)
5. Willing and capable of interacting with the informed consent process

Exclusion Criteria:

1. Unwillingness or inability to complete any of the major aspects of the study protocol, including magnetic resonance imaging (i.e., due to claustrophobia), drug cue rating, or behavioral assessment.
2. Abstinence from methamphetamine for more than 6 months based on self-report
3. Schizophrenia or bipolar disorder based on the MINI interview
4. Active suicidal ideation with intent or plan determined by self-report or assessment by PI or study staff during the initial screening or any other phase of the study
5. Positive drug test for amphetamines, opioids, cannabis, alcohol,Phencyclidine (PCP), or cocaine confirmed by breath analyzer and urine tests
6. Any active skin disorder that affects skin integrity of the scalp
7. Having any condition that would preclude undergoing an fMRI scan or tDCS stimulation based on the fMRI safety and tDCS safety checklists
8. Unstable medical disorder reported in subject's medical history or by a clinician assessment
9. History of seizure
10. Non-correctable vision or hearing problems.
11. Any other condition the PI or study staff feel would put the subject at risk for entering the study

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2017-11-30 (Actual); Primary Completion 2019-02-10 (Actual); Study Completion 2019-02-10 (Actual)

PRIMARY OUTCOMES:
Change in Drug Cue Reactivity BOLD Signal in fMRI from before to after Intervention | Immediate before and immediate after intervention
  Drug Cue Reactivity BOLD Signal is measured as average blood oxygen level dependent (BOLD) signal difference with voxel-wise analysis in the regions of interests (ROIs) (prefrontal cortex parcels, insula segments, striatum nuclei, thalamus nuclei and extended amygdala nuclei) in craving > neutral contrast in drug cue exposure fMRI task with blocks of neutral and drug related images
Change in Drug Cue Reactivity Self-Report from before to after Intervention | Immediate before and immediate after intervention
  Drug cue reactivity self-report is measured as the difference in subjective response to "On a scale of 0-100, How much drug craving are you experiencing RIGHT NOW" measured on a visual analog scale (0-100) before and after drug cue exposure fMRI task

SECONDARY OUTCOMES:
Change in Cortical-Subcortical Connectivity in Resting State fMRI from before to after Intervention | Immediate before and immediate after intervention
  Cortical-Subcortical Connectivity is measured as correlation between resting-state average blood oxygen level dependent (BOLD) signal time series in subcortical ROIs and voxels within prefrontal cortex and Insula
Change in Cortical-Subcortical Task-based Connectivity in Cue Exposure fMRI from before to after Intervention | Immediate before and immediate after intervention
  Cortical-subcortical task-based connectivity in cue exposure fMRI is measured as psychophysiological interaction (PPI) between average blood oxygen level dependent (BOLD) signal time series in subcortical ROIs and voxels within prefrontal cortex and insula, using craving > neutral contrast regressor
Change in RAI in Resting State fMRI from before to after Intervention | Immediate before and immediate after intervention
  Resource Allocation Index (RAI) is measured with the correlation among default mode network (DMN), saliency network (SN) and Executive Control Network (ECN) in resting state fMRI based on Lerman, et al., 2014.
Change in Area Under Electrode Connectivity in Resting State fMRI from before to after Intervention | Immediate before and immediate after intervention
  Area under electrode connectivity is measured with voxel-wise correlation between average blood oxygen level dependent (BOLD) signal in the cortical area under the Anode and Cathode electrodes and whole brain
Change in Area Under Electrode Task-based Connectivity in Cue Exposure fMRI from before to after Intervention | Immediate before and immediate after intervention
  Area under electrode task-based connectivity is measured with voxel-wise Psychophysiological Interaction (PPI) between average blood oxygen level dependent (BOLD) signal in the cortical area under the Anode and Cathode electrodes and whole brain using craving > neutral contrast regressor in block-design drug cue exposure fMRI task
Change in Momentary Craving Self-Report from before to after Intervention | Immediate before and immediate after intervention
  Momentary craving self-report is assessed with subjective response to "On a scale of 0-100, How much drug craving are you experiencing RIGHT NOW" measured on a visual analog scale (0-100)

OTHER OUTCOMES:
Change in Drug Cue Control Response from before to after Intervention | Immediate before and immediate after intervention
  Drug cue control response is measured as the difference in subjective response to "On a scale of 0-100, How much CONTROL over your drug craving are you experiencing RIGHT NOW" measured on a visual analog scale (0-100) before and after drug cue exposure fMRI task
Change in DI DDQ Score from before to after Intervention | Immediate before and immediate after intervention
  DI DDQ score is measured as response to the "desire and intention" (DI) subscore of the Desire for Drug Questionnaire (DDQ) for Methamphetamine (Franken, et al., 2002).
Change in NR DDQ Score from before to after Intervention | Immediate before and immediate after intervention
  NR DDQ score is measured as response to the "negative reinforcement" (NR) subscore of the Desire for Drug Questionnaire (DDQ) for Methamphetamine (Franken, et al., 2002).
Change in DDT Score from before to after Intervention | Immediate before and immediate after intervention
  DDT score is measured with responses to the Delayed Discounting Task (DDT) (Green & Myerson, 2004)

CONTACTS AND LOCATIONS:
Overall Officials: Hamed Ekhtiari, MD, PhD, Principal Investigator — Laureate Institute for Brain Research
Locations (1):
- Laureate Institute for Brain Research, Tulsa, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: No